CLINICAL TRIAL: NCT02342626
Title: CDC SIP: Rochester Prevention Research Center: Development and Evaluation of an Active Surveillance Decision Aid for Men With Low or Intermediate Grade Prostate Cancer
Brief Title: Devel. and Eval. of an Active Surveillance Decision Aid for Men With Low or Intermediate Grade Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, James Dolan, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS14115
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Adenocarcinoma of Prostate
Keywords: Prostate; Cancer; Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma | interventions — Dashboard Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No use of the decision aid dashboard before, during or after the treatment decision time period.
- Dashboard (Experimental): Use of the decision aid dashboard before, during and after the treatment decision time period.
  Interventions: Behavioral: Dashboard

INTERVENTIONS:
Behavioral: Dashboard — With the health care provider, subjects will use the decision dashboard to augment the discussion of treatment options.
  Arms: Dashboard

SUMMARY:
The overall goal of this project is to test an interactive, multi-media decision aid in the form of an electronic clinical decision dashboard designed to improve the quality of clinical decision making for initial treatment of patients with newly diagnosed, low or intermediate risk prostate cancer.

DETAILED DESCRIPTION:
The overall goal of this project is to test an interactive, multi-media decision aid in the form of an electronic clinical decision dashboard designed to improve the quality of clinical decision making for initial treatment of patients with newly diagnosed, low or intermediate risk prostate cancer.

Specifically, we propose to conduct a clinical trial to compare the effects of a prostate decision dashboard versus usual care on:

1. patient knowledge regarding the treatment options available for low or intermediate risk prostate cancer,
2. measures of the decision making process including decisional conflict and the extent to which decisions were made via a shared decision making process,
3. the treatments selected, and
4. 3-6 and 9-12 month outcome assessments of clinical status, decision regret, cancer-related quality of life including worry, functional status, and treatment side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 85 years
* Sex: male
* Race/ethnicity: no restrictions
* Diagnosis: Patients will be eligible for the study if they have not yet decided on a management plan and present with either:
* localized, low grade prostate cancer, defined as Gleason score ≤ 6, T1-T2a stage cancers, and PSA values < 10 ng/ml, OR
* Intermediate risk prostate cancer, defined as Gleason score = 7, T2b-T2c stage cancers (these tumors involve more of the prostate but do not extend beyond the prostatic capsule), or PSA 10-20 ng/ml
* Willing to participate and able to give informed consent
* Able to adequately see the study intervention which is an interactive decision dashboard & complete study-related questionnaires
* Able to understand English language adequately to use the decision dashboard and complete study-related questionnaires

Exclusion Criteria:

* Unable to complete study-related tasks due to cognitive deficits or English non-fluency
* Unwilling to participate.
* Deemed clinically unsuitable for active surveillance as a prostate cancer management option

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Increase in KUJ score through education | 2 years
  The use of the dashboard will increase patient knowledge and understanding of treatment options as measured using KUJ questionnaire.

SECONDARY OUTCOMES:
Measure of overall quality and satisfaction with initial treatment decision. | 2 years
  The use of the dashboard will improve the overall quality and satisfaction with initial treatment decisions as measured by a) decisional conflict, b) patient quality of life, and c) post-decision regret, using the PORPUS questionnaire and Decisional Regret questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: James G Dolan, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No